CLINICAL TRIAL: NCT04832607
Title: Treatment of Chemo-refractory Viral Infections After Allogeneic Stem Cell Transplantation With Multispecific T Cells Against CMV, EBV and AdV: A Phase III, Prospective, Multicentre Clinical Trial
Brief Title: Multivirus-specific T-cell Transfer Post SCT vs AdV, CMV and EBV Infections
Acronym: TRACE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tobias Feuchtinger (Other)
Collaborators: European Commission (Other); Simbec-Orion Group Ltd, Merthyr Tydfil, UK (Unknown); Miltenyi Biotec B.V. & Co. KG, Bergisch Gladbach, Germany (Unknown); Leiden University Medical Center, LUMC, Leiden, The Netherlands (Unknown); Central Hospital, Nancy, France (Other); University Hospital, Ghent (Other); Ospedale Pediatrico Bambino Gesù, OPBG, Rome, Italy (Unknown); Newcastle University, UNEW, Newcastle, UK (Unknown); Vall d'Hebron Institute of Oncology (Other)
Responsible Party: Sponsor-Investigator, Tobias Feuchtinger, Prof. Dr. med Tobias Feuchtinger, University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRACE; 2018-000853-29 (EudraCT Number); DRKS00018985 (Other: Deutsches Register Klinischer Studien)
Record Dates: First submitted 2021-03-19; First posted 2021-04-06 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: AdV Infection; EBV Infection; CMV Infection; Stem Cell Transplant Complications
MeSH Terms: conditions — Adenoviridae Infections; Epstein-Barr Virus Infections; Cytomegalovirus Infections

STUDY DESIGN:
Intervention Model Description: 2 (verum): 1 (Placebo) randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be stratified with respect to three age groups: Children up to 6 years, children >6 and up to 18 years, and adults >18 years. Accordingly, for each stratum, a separate randomization list will be provided. Randomization will be performed by a representative of the Simbec-Orion Group who will be independent in the sense that he / she will otherwise not be involved in the TRACE trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multivirus (CMV, EBV, AdV)-specific T cells (Experimental): Allogeneic CD4+ and CD8+ T lymphocytes ex vivo incubated with synthetic peptides of the viral antigens of Cytomegalovirus, Adenovirus and Epstein-Barr Virus
  Max dose:
  * HLA-matched (8/8) donors: 1.0 x 10e5 T cells/kg recipient BW
  * HLA-mismatched donors: 2.5 x 10e4 T cells/kg recipient BW
  Min. dose:
  - 10 T cells/kg recipient BW
  Interventions: Other: Multivirus (CMV, EBV, AdV)-specific T cells
- Sodium chloride (Placebo Comparator): Suspension of multivirus-specific T cells in 20 mL of 0.9% NaCl + 0.5% HSA
  Interventions: Other: Multivirus (CMV, EBV, AdV)-specific T cells

INTERVENTIONS:
Other: Multivirus (CMV, EBV, AdV)-specific T cells — Cell therapy product which is individually produced for each patient and administered via IV bolus injection.

SUMMARY:
Haematopoietic stem cell transplantation (HSCT) can expose patients to a transient but marked immunosuppression, during which viral infections are an important cause of morbidity and mortality. Adoptive transfer of virus-specific T cells is an attractive approach to restore protective T-cell immunity in patients with refractory viral infections after allogeneic HSCT. The aim of this Phase III trial is to confirm efficacy of this treatment in children and adults.

DETAILED DESCRIPTION:
For a growing number of patients suffering from various conditions as, e.g., haematological malignancies or diverse genetic disorders, haematopoietic stem cell transplantation (HSCT) or bone marrow transplantation offer the only possible curative options. However, HSCT is associated with three major risks: graft rejection, graft-versus-host disease (GvHD) and opportunistic, mostly viral, infections or reactivations resulting from delayed immune reconstitution. Delayed immune reconstitution, however, often is the direct result of the severe pre-transplantation conditioning treatment and T-cell depletion of the transplant necessary to fight the risks of graft rejection and GvHD. Therefore, the risk for life-threatening opportunistic, mostly viral, infections is increased in post-transplantation patients. The most common infections after HSCT are Cytomegalovirus (CMV), Epstein-Barr virus (EBV) and Adenovirus (AdV).

The standard treatment approach for viral infections/reactivations is chemotherapy which shows limited efficacy and does not restore immunity. Therefore, effective new treatment options are required for this condition.

Previous investigations have shown that sufficient T-cell immunity is essential for the control and prevention of viral reactivations and newly occurring infections after HSCT. The infusion of T-cells is therefore a promising new approach to treat immune-comprised patients. However, infusion with unselected T cells is associated with an increased risk for GvHD due to the high content of alloreactive T cells. A very promising approach to minimize this problem is to remove alloreactive T cells and enrich, isolate and purify virus-specific T cells.

This approach has been studied for nearly two decades and the data published up to date indicate that virus-specific T-cell responses after adoptive T-cell transfer protect against virus-related complications post HSCT and restore T-cell immunity, in particular for AdV-, CMV- and EBV-infections. Despite these promising results, virus-specific T-cell transfer is not yet translated into daily clinical practice due to the lack of prospective clinical trials confirming the efficacy of this treatment approach.

The overall goal of this Phase III, double-blind placebo-controlled study is to test efficacy of multivirus-specific T cells to bring this treatment method in clinical routine. Multivirus-specific T cells generated in this study will be directed against all three most common post-HSCT viral infections: AdV, CMV and EBV. Thus, T-cell immunity will be restored to fight and prevent new viral infections.

After an initial screening visit, patients eligible to participate in the study will be treated within 28 days after screening. Patients will be randomized in a 2:1 (treatment: placebo) ratio and receive a single infusion with either multivirus-specific T cells or placebo. Patients will be followed up on the day of treatment, 1 day after and 1, 2, 4, 8 and 15 weeks after treatment. Treatment success will be measured by assessing different parameters including symptoms, quality of life, viral load and T-cell immunity in blood samples.

Patients eligible to participate in this study are adult and paediatric patients who have received allogeneic stem cell transplantation and suffer from new or reactivated EBV, AdV or CMV infection refractory to standard antiviral treatment for two weeks. Patients from the six European countries Germany, Belgium, Netherlands, UK, France and Italy will be enrolled. In total 130 patients plus 19 screening failures are expected to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult or paediatric patients (> 2 months of age) after allogeneic stem cell transplantation (SCT) (no time restrictions apply) suffering from new or reactivated CMV or EBV or AdV infection refractory to standard antiviral treatment for two weeks (defined as no decrease or insignificant decrease of less than 1log in viral load over two weeks) as confirmed by quantitative blood PCR analysis.
2. Original HSCT-donor available with an immune response at least to the virus causing the therapy-refractory (=underlying) infection.
3. Written informed consent given (patient or legal representative) prior to any study-related procedures.

Exclusion Criteria:

1. Patient with acute GvHD > grade II or extensive chronic GvHD at the time of IMP transfer
2. Patient receiving steroids (>1 mg/kg BW Prednisone equivalent) at Screening.
3. Therapeutic donor lymphocyte infusion (DLI) from 4 weeks prior to IMP infusion until 8 weeks post IMP infusion. Prescheduled prophylactic DLI ≤3x105 T cells/kg BW in case of T-cell depleted HSCT is not considered an exclusion criterion.
4. Patient with organ dysfunction or failure as determined by Karnofsky (patients >16 years) or Lansky (patients ≤16 years) score ≤30%
5. Concomitant enrolment in another clinical trial interfering with the endpoints of this study
6. Any medical condition which could compromise participation in the study according to the investigator's assessment
7. Progression of underlying disease (disease that has led to the indication of HSCT, e.g. leukaemia) that will limit the life expectance below the duration of the study
8. Second line or experimental antiviral treatment other than Ganciclovir/Valganciclovir, Foscarnet, Cidofovir and Rituximab until 8 weeks after IMP Infusion or prophylactic Treatment other than Aciclovir or Letermovir throughout the study except approved by sponsor
9. Known HIV infection. In case patients do not have a negative HIV test performed within 6 months before enrolment in the study, HIV negativity has to be confirmed by a negative laboratory test.
10. Female patient who is pregnant or breast-feeding. Female patient of child-bearing potential (i.e. post menarche and not surgically sterilized) or male patient of reproductive potential not willing to use an effective method of birth control from Screening until the last follow-up visit (FU6, Visit 8).

    Note: Women of childbearing potential must have a negative serum pregnancy test at study entry ≤7 days before IMP administration on Day 0. Acceptable birth control methods are hormonal oral contraceptive ('pill'), contraceptive injection or patch, intrauterine pessar or the combination of two barrier methods. The combination of female and male condomes is NOT acceptable. If the male partner is sterilized, no further contraceptive is required. Women of post-menopausal status (no menses for 12 months without an alternative medical cause) are also not required to use contraceptives during the study.
11. Known hypersensitivity to iron dextran
12. Patients unwilling or unable to comply with the protocol or unable to give informed consent.

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2019-08-27 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Viral clearance | 8 weeks after treatment
  Percentage of patients with viral clearance (defined as two consecutive negative PCRs) to determine efficacy of multispecific T-cell transfer in patients with chemo-refractory viral infections after allogeneic stem cell transplantation
Disease Progression | day 7 until week 8 after treatment
  Percentage of patients with progression between Day 7 and Week 8 after T-cell Transfer to determine efficacy of multispecific T-cell transfer in patients with chemo-refractory viral infections after allogeneic stem cell transplantation

SECONDARY OUTCOMES:
Incidence of acute GvHD | 15 weeks after treatment
  Incidence of newly occurring acute GvHD grade I from Day 0 to Week 8 and Week 15.
Incidence of chronic GvHD | 15 weeks after treatment
  Incidence of chronic GvHD from Day 7 to Week 8 and to Week 15 after treatment.
Time to newly occuring GvHD | 15 weeks after treatment
  Time to newly occurring acute and chronic GvHD.
Severity of GvHD | week 8 and 15 week after treatment
  Severity of acute GvHD ≥ grade II until Week 8 and Week 15.
Incidence of acute toxicity | 15 minutes, 30 minutes, 2 hours and 4 hours post T-cell/placebo transfer
  Acute maximum toxicity on the day of T-cell transfer evaluated by measuring vital signs prior to and at different times after the T-cell transfer from 1 hour prior to T-cell transfer to 4 hours post infusion.
Severity of acute toxicity | 15 minutes, 30 minutes, 2 hours and 4 hours post T-cell/placebo transfer
  Monitoring of adverse events infusion.
Change in viral load of underlying viral infection | 8 weeks after treatment
  Change in viral load of underlying viral infection as assessed by quantitative PCR analysis of peripheral blood; samples taken weekly from Day 7 to Week 8 after IMP transfer as compared to samples taken at Day 0.
Time to viral load change of underlying viral infection | 15 weeks after treatment
  Time to 1 log change in viral load.
Percentage of viral decrease | 8 weeks after treatment
  Percentage of patients with ≥1 log decrease in CMV, EBV or AdV viral load at Week 8.
Viral reactivations | 15 weeks after treatment
  Number of reactivations of the underlying viral infection following initial viral clearance until end of follow-up.
Clinical response/resolution of symptoms of underlying viral infection | 8 weeks after treatment
  Number of patients with reduction or clearance of clinical symptoms of underlyingviral infection from Day 7 to Week 8 after IMP transfer as compared to Day 0.
Overall survival | 15 weeks after treatment
  Overall survival rate (OS): From Day 0 to end of follow-up.
Necessity of antiviral chemotherapy | Day 7 until Week 8
  Number of days requiring antiviral chemotherapy after T-cell transfer from Day 7 to Week 8 after T-cell transfer.
Duration of antiviral chemotherapy | 8 weeks after treatment
  Time to last administration of defined antiviral medication or switch to prophylactic treatment from Day 0 to Week 8 after IMP transfer.
Incidence of viral infections other than underlying viral infection | 15 weeks
  Number of new viral reactivations (CMV, AdV or EBV) other than the underlying viral infection per patient as assessed by PCR analysis and clinical symptoms throughout the study to evaluate the putative prophylactic effect of the treatment.
Days of hospitalization | 8 weeks
  Number of days hospitalized after IMP transfer from Day 7 to Week 8.
Life quality in adults | Screening and Week 8.
  EQ-5D for adult patients (≥18 years) at Screening and Week 8 to evaluate life quality in adults. A scale from 0 to 100 is used with 100 being best value and 0 the worst.
Life quality in adults | Screening and Week 8
  FACT-BMT for adult patients (≥18 years) at Screening and Week 8 to evaluate life quality in adults.
  The patients have to answer questions about their physicial, social, emotional and functional wellbeing. A scale from 0 to 4 is used with 0= not at all, 1= a little bit, 2=somewhat, 3=quite a bit, 4=very much.
Life quality in children | Screening and Week 8
  PEDS-QL for paediatric patients (<18 years) at Screening and Week 8 to evaluate life quality in children.
  The patients and /or their parents have to answer questions about pain and hurt, fatigue and sleep, nausea, worry, Nutrition, thinking and communication.
  A scale from 0 to 4 is used with 0=never a Problem, 1=almost never a problem, 2= sometimes a problem, 3=often a problem, 4= almost always a problem.
Effect on the patient's T-cell phenotype in vivo | Screening until Week 15
  T-cell phenotyping, samples taken at Screening, Day 0 and each visit from Day 7 to Week 15 after treatment.
Effect on the patient's number of expanded T cells | Screening until Week 15
  Analysis of virus-specific T cells: frequencies of in vivo expanded virus-specific T cells in peripheral blood samples taken at Screening, Day 0, Day 7 to Week 15 after treatment.
Quality of the IMP and performance of the CliniMACS® Prodigy | Before IMP release (between Screening and Day 0)
  Assessment of the cellular composition, in particular the percentage of IFN-gamma+ cells, in the IMP.
Evaluation of the drop-out rate | at Day 0 (planned treatment day)
  Drop-out rate at Day 0 and reasons for drop-out.
Time from inclusion to administration of the IMP | Screening until Day 0 (treatment day)
  Number of days from Screening to Day 0 (day of IMP transfer) to evaluate the required time frame.
Adverse events | 15 weeks
  Documentation of incidence, severity and type of adverse events from Day 0 to Week 8 and serious adverse events throughout the study to evaluate safety.
Physical examination | Screening to Week 8
  Physical examinations will be conducted to identify possible clinically significant pathologies. These findings will be recorded at each visit. The Karnofsky/Lansky index will be included in the physical examination at Screening and at Week 8 only.
Vital Sign - blood pressure | Screening to Week 8
  supine systolic and diastolic blood preasure in mm Hg
Vital Signs - heart rate | Screening to Week 8
  The resting heart rate in beats/min
Vital Signs - body temperature | Screening to Week 8
  Body temperature in °C (aural)
Vital Signs - body weight | Screening to Week 8
  body weight in kg
Vital Signs - respiratory rate | Screening to Week 8
  respiratory rate in breaths/min.
Incidence of abnormal laboratory values | Screening to Week 8
  haemoglobin, leukocytes, thrombocytes, dirfferential blood count (neutrophil granulocytes, lymphocytes, monocytes and easinophil granulocytes), total and conjugated Bilirubin, C reactive Protein (CRP), creatinine, Alanin aminotransferase (ALT), Aspartate aminotransferase (AST), Gamma glutamyl Transferase (GGT), Lactate Dehydrase (LDH), Urea.
  A list of normal ranges will be provided from each site.
Concomitant medication until Week 8 | 8 weeks after treatment
  All concomitant medication will be recorded from Screening until Week 8. The generic name, indication, route of administration, dose/ unit, start and stop date or ongoing, way of application will be documented.
Concomitant medication until Week 15 | 15 weeks after treatment
  During follow-up Week 15, only antiviral therapy, immunosuppression and SAE-related concomitant medication as well as chemotherapy will be documented.
  The generic name, indication, route of administration, dose/ unit, start and stop date or ongoing, way of application will be documented.
  Cellular treatment also has to be documented as concomitant medication.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Feuchtinger, Prof, Principal Investigator — Medical Center - University of Freiburg
Locations (33):
- Belgium (5):
  - Institut Jules Bordet (JBI), Brussels
  - UZ Brussel, Brussels
  - Ghent Universal Hospital (UZG), Ghent
  - UZ Leuven, Leuven
  - Université de Liège (ULG), Liège
- France (6):
  - Hôpital Jeanne de Flandre, CHU Lille, Lille
  - Institut d'Hématologie et Oncologie Pédiatrique (IHOPe), Lyon
  - Centre Hospitalier Régional Universitaire de Nancy (CHRU), Nancy
  - Hôpital de la Pitie-Salpêtrière, Paris
  - Hôpital Necker - Enfants Malades, Paris
  - Hôpital Robert Debré, Paris
- Germany (15):
  - Charité Berlin (Campus Virchow-Klinikum) - Klinik für Pädiatrie mit Schwerpunkt Onkologie und Hämatologie, Berlin
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Düsseldorf - Klinik für Kinder-Onkologie, -Hämatologie und klinische Immunologie, Düsseldorf
  - Universitätsklinikum Essen - Pädiatrische Hämatologie-Onkologie, Essen
  - Universitätsklinikum Freiburg - Klinik für Pädiatrische Hämatologie und Onkologie, Freiburg im Breisgau
  - Medizinische Hochschule Hannover - Zentrum für Kinderheilkunde und Jugendmedizin, Hanover
  - Universitäsklinikum Leipzig - Medizinische Klinik und Poliklinik I, Leipzig
  - LMU Klinikum - Dr. v. Haunersches Kinderspital, Munich
  - Klinikum rechts der Isar der Technischen Universität - Kinderklinik Schwabing, Munich
  - LMU Klinikum - Medizinische Klinik und Poliklinik III, München
  - Klinikum rechts der Isar der Technischen Universität - Klinik und Poliklinik für Innere Medizin III, München
  - Universitätsklinikum Regensburg - Pädiatrische Hämatologie, Onkologie und Stammzelltransplantation, Regensburg
  - Universitätsklinikum Tübingen, Center for Pediatric Clinical Studies (CPCS), Tübingen
  - Universitätsklinikum Würzburg - Medizinische Klinik und Poliklinik II & Zentrum Innere Medizin (ZIM), Würzburg
  - Universitätsklinikum Würzburg - Pädiatrische Hämatologie, Onkologie und Stammzelltransplantation, Würzburg
- Italy (2):
  - Ospedale Pediatrico Bambino Gesù (OPBG), Rome
  - Ospedale Infantile Regina Margherita - Oncoematologie Pediatrica, Turin
- Leiden University Medical Centre (LUMC) - Department of Hematology, Leiden, Netherlands
- Spain (4):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitario Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No